CLINICAL TRIAL: NCT02154113
Title: Baseline Controlled Two-arm Multi-Center Study to Evaluate the Safety and Efficacy of Combined Multi-Focus Treatments of UltraShape® Contour I V3 System and VelaShape II Device for Non-Invasive Circumference Reduction
Brief Title: Ultrashape System in Combination With VelaShape II Device for Circumferential Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US-CA 02
Record Dates: First submitted 2014-05-27; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Abdominal Fat
Keywords: Syneron; Velashape; ELOS; Ultrashape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Velashape II device (Active Comparator): Controlled infrared (IR) light and conducted bipolar radiofrequency (RF) energies with mechanical manipulation.
  Interventions: Device: Velashape II
- Ultrashape (Active Comparator): The UltraShape Contour I V3 uses focused ultrasound to produce localized mechanical motion within fat tissues and cells for the purpose of producing mechanical cellular membrane disruption.
  Interventions: Device: Ultrashape

INTERVENTIONS:
Device: Ultrashape — All subjects receive 3 successive Ultrashape treatments every two weeks in the anterior abdomen.
  Arms: Ultrashape
Device: Velashape II — All subjects receive 3 successive Velashape treatments every two weeks in the anterior abdomen.
  Other Names: Vela, Velashape
  Arms: Velashape II device

SUMMARY:
The purpose of this study is to compare the clinical performance of the Ultrashape system with VelaShape II device for reduction of the waist.

DETAILED DESCRIPTION:
UltraShape® Contour I V3 system is a non-invasive (not breaking the skin) focused ultrasound for body contouring purposesdesigned to selectively disrupt sub-dermal fat cells employing focused ultrasound. All other types of tissue, such as blood vessels, muscles and peripheral nerves, remain intact. There are no thermal effects. Fat-cell destruction is achieved by ultrasound-induced mechanical effects during a very short exposure time.

VelaShape is a non-invasive device for Body Reshaping and Cellulite Treatment. VelaShape combines controlled infrared (IR) light and conducted bipolar radiofrequency (RF) energies with mechanical manipulation.

ELIGIBILITY:
Inclusion Criteria:

1. Fat thickness of at least 1.5 cm in the anterior abdominal and flanks prior to initial treatment (measurement by caliper)
2. For women of child-bearing potential: negative pregnancy test in the 24 hour period prior to enrollment and 24 hour period prior to each treatment or FU visit (measured in urine)
3. General good health confirmed by medical history and skin examination of the treated area
4. Written informed consent to participate in the study
5. Ability to comply with the requirements of the study
6. BMI≤ 30

Exclusion Criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
2. Current hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease or malignancy
3. Previous liposuction in the treatment areas
4. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
5. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
6. Poor skin quality (i.e., laxity)
7. Abdominal wall diastasis or hernia on physical examination
8. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
9. Obesity (BMI > 30)
10. Childbirth within the last 12 months or women who suckling a child
11. Any acute or chronic condition which, in the opinion of the Investigator, could interfere with the conduct of the study
12. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months)
13. Inability to comply with circumference measurement procedure (e.g., inability to held breath for the required duration)
14. Participation in another clinical study
15. Previous body contouring treatments in the treatment areas

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Difference in circumference reduction between baseline and follow-up visits | Base line, 2 and 12 weeks post last treatment
  The primary efficacy endpoint in this trial is the statistical difference in circumference reduction between Control (baseline measurement, Vist 2 / Day 0) and two points of follow-up measurement: 2 weeks (Visit 5 / Day 42) and 12 weeks (Visit 8 / Day 112) following the last Tx session. The following procedure will be used to compute the Circumference Difference primary endpoint:

SECONDARY OUTCOMES:
Adverse Events | The duration of the study, an expected average of 5 months.
  Safety will be evaluated based on the incidence and severity of adverse events caused by the treatments

OTHER OUTCOMES:
Subject Satisfaction Scores | 2, 4, 6, 8,10 and 12 week in a study.
  Subject Satisfaction Scores using the Global Aesthetic Improvement (GAI) Scale at each treatment and follow-up time point post treatment: 2 week, 4 week, 6 week, 8 week, 10 week and 12 week in a study.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Mann, Study Director — Syneron Medical Ltd.
Locations (2):
- Canada (2):
  - BC Laser & SkinCare Clinic, Surrey, British Columbia
  - Cosmedica, Pointe-Claire, Quebec